CLINICAL TRIAL: NCT01986868
Title: Identification of Adverse Plaque Characteristics by Coronary Magnetic Resonance Angiography
Brief Title: Identification of Adverse Plaque Characteristics by Coronary MR Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Daniel S. Berman, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 27850
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Magnetic Resonance Angiography; CMRA; MRI with contrast; MultiHance; Optimark; Gadolinium-based contrast; MRA; MR angiography
MeSH Terms: conditions — Coronary Artery Disease | interventions — Magnetic Resonance Spectroscopy; Contrast Media; gadobenic acid; gadoversetamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Coronary MR Angiography (CMRA) (Other): Coronary MR Angiography(CMRA). A gadolinium-based contrast (Optimark or MultiHance) will be administered as well as a beta blocker which will be assigned based upon heart rate.
  Interventions: Other: Coronary MR Angiography (CMRA)

INTERVENTIONS:
Other: Coronary MR Angiography (CMRA) — Stable patients who have undergone a clinically indicated CCTA study for suspected Coronary Artery Disease will undergo a research CMRA with contrast (Multihance or Optimark)total dose of up to 0.2 mmol/kg IV. Possible administration of oral beta-blocker (metoprolol)intravenous doses of 5mg IV metoprolol may be given every 2 minutes up to a maximal dose of 15 mg IV.
  Other Names: MRI with contrast; MultiHance; Optimark; Gadolinium-based contrast; MRA; MR Imaging; MR angiography

SUMMARY:
This is a pilot study to determine whether coronary magnetic resonance angiography(CMRA)can identify adverse plaque characteristics (buildup of fat, cholesterol, calcium, and other substances found in the blood) seen on coronary computed tomography angiography(CCTA) and evaluate whether there is a relationship between the adverse plaque characteristics and the presence of coronary artery wall inflammation.

DETAILED DESCRIPTION:
This pilot study will examine 20 stable patients who have undergone a clinically-indicated coronary computed tomography angiography (CCTA) for suspected Coronary Artery Disease. They will be invited to undergo a research coronary Magnetic Resonance Imaging scan with contrast(CMRA). Based upon the subject's heart rate, a beta blocker may be administered as its use has been shown to be effective in producing better images as it widens the arteries.

Researchers will use newly developed non-invasive coronary MRA techniques to compare information shown on the research CMRA with the clinical CCTA. While CCTA has been demonstrated to be able to provide data on adverse plaque characteristics (APC's), the ability of CMRA to evaluate these features is not established.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Ability to comprehend and sign informed consent
* Presence of a non-calcified or mixed plaque without high-grade stenosis in the left main or a proximal coronary artery segment AND at least one APC present in this plaque by CCTA (defined as LAP with <30 Hounsfield units or PR with ≥10% increase in the maximal vessel diameter within the plaque as compared to a proximal reference segment as previously described10).

Exclusion Criteria:

* High-grade stenosis (≥50% stenosis of the left main artery or ≥70% stenosis of another proximal coronary segment);
* Coronary artery stent in the segment with the reference plaque
* Possible pregnancy
* Glomerular filtration rate <45 ml/min
* More than 90 days between CCTA and CMRA study
* Any significant arrhythmia (e.g. atrial fibrillation, frequent ectopy)
* Significant asthma
* History of 2nd or 3rd degree heart block
* Allergy or known intolerance to beta-blockers
* Use of phosphodiesterase inhibitor (e.g. Viagra) within the last 48 hours
* Rapid heart rate (heart rate ≥90 beats/minute)
* Severe aortic stenosis (Aortic valve area <1.0 cm2 or mean gradient >30 mmHg)
* Systolic blood pressure <100 mmHg
* Other contraindication to MRI, including metallic implants (valve replacement, pacemaker, implantable cardiac defibrillator, metallic spine material), intracranial clips, metallic fragments in eyes, and claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2018-01-24 (Actual)

PRIMARY OUTCOMES:
Adverse plaque characteristics present on CMRA | one day

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Berman, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States